CLINICAL TRIAL: NCT06288113
Title: Re-Treatment With 177Lu-PSMA-617 Molecular Radiotherapy for Metastatic Castration Resistant Prostate Cancer: A Prospective Phase 2 Trial (RE-LuPSMA STUDY)
Brief Title: Re-treatment With 177Lu-PSMA-617 for the Treatment of Metastatic Castration-Resistant Prostate Cancer, RE-LuPSMA Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-001509; NCI-2024-00310 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-001509 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2024-02-05; First posted 2024-03-01 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Castration-Resistant Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Pluvicto; Magnetic Resonance Spectroscopy; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (177Lu-PSMA-617) (Experimental): Patients receive 177Lu-PSMA-617 IV on day 1 of each cycle. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive gallium Ga 68 gozetotide IV and undergo PET/CT at screening and on study, undergo SPECT/CT on study, and undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Gallium Ga 68 Gozetotide; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT and SPECT/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Other: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; AAA 517; AAA-517; AAA517; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Drug: Lutetium Lu 177 Vipivotide Tetraxetan — Given IV
  Other Names: 177Lu-labeled PSMA-617; 177Lu-PSMA-617; AAA 617; AAA-617; AAA617; Lu177-PSMA-617; Lutetium Lu 177-PSMA-617; LUTETIUM LU-177 VIPIVOTIDE TETRAXETAN; Lutetium-177-PSMA-617; Pluvicto
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
This phase II trial tests how well re-treatment with 177Lu-PSMA-617 works in treating patients with prostate cancer that has spread from where it first started (primary site) to other places in the body (metastatic), that continues to grow or spread after the surgical removal of the testes or medical treatment to block androgen production (castration-resistant), and that has shown a favorable response to initial treatment with 177Lu-PSMA-617. 177Lu-PSMA-617 is a radioactive drug. It binds to a protein called prostate specific membrane antigen (PSMA), which is expressed by some types of prostate tumor cells. When 177Lu-PSMA-617 binds to PSMA-expressing tumor cells, it delivers radiation to the cells, which may kill them. Re-treatment with 177Lu-PSMA-617 in patients who had a favorable response to initial 177Lu-PSMA-617 treatment may improve survival outcomes and disease response in patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the treatment efficacy of re-challenge lutetium Lu 177 vipivotide tetraxetan (177Lu-PSMA-617) therapy (for a maximum of 6 additional cycles) in patients with metastatic castration-resistant prostate cancer (mCRPC) who had a favorable response to a prior regimen of 177Lu-PSMA-617 therapy.

SECONDARY OBJECTIVES:

I. To determine the safety of re-challenge 177Lu-PSMA-617 therapy by Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

II. To determine the rate of patients who have a prostate-specific antigen (PSA) response (defined as a PSA decline of ≥ 50% during re-challenge 177Lu-PSMA-617 therapy).

III. To determine biochemical progression-free survival (PFS) according to Prostate Cancer Working Group 3 (PCWG3) guidelines.

IV. To determine overall survival (OS) from the start (cycle 1 day 1) of the first regimen of 177Lu-PSMA-617 therapy.

V. To determine OS from the end (day 1 of the final cycle) of the first regimen of 177Lu-PSMA-617 therapy.

VI. To determine radiographic progression-free survival (rPFS) according to Response Evaluation Criteria in PSMA positron emission tomography (PET)/computed tomography (CT) (RECIP) criteria.

VII. To determine the impact of re-challenge 177Lu-PSMA-617 therapy on bone pain level, health-related quality of life, and performance status (Eastern Cooperative Oncology Group [ECOG]) using established standardized questionnaires.

EXPLORATORY OBJECTIVE:

I. To determine the dosimetry in organs and tumor lesions of re-challenge 177Lu-PSMA-617 therapy using a 24-hour single-time-point dosimetry protocol.

OUTLINE:

Patients receive 177Lu-PSMA-617 intravenously (IV) on day 1 of each cycle. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive gallium Ga 68 gozetotide IV and undergo PET/CT at screening and on study, undergo single photon emission computed tomography (SPECT)/CT on study, and undergo collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up within 8 weeks of their last treatment cycle and then every 3 months for up to a total of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have mCRPC
* Patients must have received at least one regimen of chemotherapy for mCRPC
* Patients must have received at least one androgen receptor signaling inhibitor (ARSI)
* Patients must have previously completed at least 4 cycles of 177Lu-PSMA-617 therapy
* Patients must have had a favorable response to the first regimen of 177Lu-PSMA-617 therapy defined as:

  * PSA decline of ≥ 50% at any time during the first regimen of 177Lu-PSMA-617 therapy AND
  * No new prostate cancer therapy within two months of completing the first regimen of 177Lu-PSMA-617 therapy (first-generation androgen deprivation therapy [ADT] is allowed). Concomitant prostate cancer therapy that was administrated during the first regimen of 177Lu-PSMA-617 therapy and continued afterwards is allowed
* Patients must have had a PSA increase after the first regimen of 177Lu-PSMA-617 therapy, confirmed by a second measurement ≥ 3 weeks apart
* Patients must meet PSMA PET/CT VISION criteria. PSMA PET/CT must have been completed within 8 weeks of the planned first cycle of re-challenge 177Lu-PSMA-617 therapy and at least 6 weeks after completion of the first regimen of 177Lu-PSMA-617 therapy
* White blood cells > 2,500 cells/µL
* Absolute neutrophil count > 1,500 cells/µL
* Hemoglobin > 9.0 g/dL
* Platelets > 100,000 cells/µL
* Patients must have the ability to understand and sign an approved informed consent form (ICF) and comply with all protocol requirements

Exclusion Criteria:

* Patient received new prostate cancer therapy within two months of completing the first regimen of 177Lu-PSMA-617 therapy (first-generation ADT (adenosine triphosphate) is allowed). This can include apalutamide, enzalutamide, abiraterone, chemotherapy, immunotherapy, radionuclide therapy, PARP inhibitor, or any biological therapy. Concomitant prostate cancer therapy that was administrated during the first regimen of 177Lu-PSMA-617 therapy and continued afterwards is allowed
* Patient received myelosuppressive therapy (including docetaxel, cabazitaxel, 223Ra, and 153Sm) or other radionuclide therapy within the last 6 weeks
* Patient with creatinine clearance < 50 mL/min

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2027-01-27 (Estimated)

PRIMARY OUTCOMES:
12-month overall survival | Assessed at 12 months
  12-month overall survival (OS) of patients with mCRPC who previously had a favorable response to a first regimen of 177Lu-PSMA-617 and are treated with re-challenge 177Lu-PSMA-617 therapy

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Assessed approximately at 2 years
  Overall and grade ≥ 3 AEs will be defined and graded according to Common Terminology Criteria for Adverse Events version 5.0. Descriptive statistics will be used to report the number and percentage of patients who experience AEs during re-challenge therapy. Separate statistics will be reported for grade ≥ 1 AEs and for grade ≥ 3 AEs. These descriptive statistics will be presented for the whole treatment as well as separately for each cycle. In addition, the relationship of AE to the study drug (related versus not related) will be reported. Results from laboratory test, physical examinations, and patient surveys will be used.
Rate of prostate specific antigen (PSA) response | Assessed approximately at 36 weeks
  Will be defined as a PSA decline of ≥ 50% during re-challenge therapy on two measurements ≥ 3 weeks apart. Descriptive statistics will be used to report the number and percentage of patients who had a PSA response to re-challenge therapy. The number and percentage of patients with any decrease in serum PSA level compared to the baseline PSA at time of study enrollment will be reported as well.
Biochemical progression-free survival (PFS) | Assessed approximately at 2 years
  Will be evaluated using Prostate Cancer Working Group 3 guidelines.
Overall Survival from start of first regimen | Assessed approximately at 2 years
  To determine OS from the start of the first regimen of 177Lu-PSMA-617 therapy (Cycle 1 Day 1) (each cycle is 6 weeks) through study completion.
Overall survival from the end of the first regimen | Assessed approximately at 2 years
  To determine OS from the end of the first regimen of 177Lu-PSMA-617 therapy (Day 1 of the final cycle) (each cycle is 6 weeks) through study completion.
Radiographic progression-free survival (rPFS) | approximately two years.
  To determine radiographic progression-free survival (rPFS) according to Response Evaluation Criteria in PSMA PET/CT (RECIP) criteria through study completion.
Bone Pain | approximately 36 weeks.
  Proportion of patients who initially had bone pain who experienced pain response with re-challenge 177Lu-PSMA-617 therapy
Changes in health-related quality of life_Functional Assessment of Cancer Therapy - Radionuclide Therapy (FACT-RNT). | approximately 36 weeks.
  The Functional Assessment of Cancer Therapy - Radionuclide Therapy (FACT-RNT) is a patient-reported outcome (PRO) tool designed to measure symptoms and toxicities among prostate cancer patients receiving radionuclide therapy (RNT). The total score can range from 0 to 60, with higher scores indicating better quality of life and fewer symptoms or side effects related to radionuclide therapy (RNT).
Changes in health-related quality of life_Brief Pain Inventory Short form | approximately 36 weeks.
  Pain response will be evaluated as at least a 2-point improvement from baseline without an overall increase in opiate use. evaluated using Brief Pain Inventory Short form (BPI-SF). The Brief Pain Inventory Short Form (BPI-SF) is a widely used tool for assessing pain severity and its impact on daily life. Ratings are on a scale from 0 (does not interfere) to 10 (completely interferes).
  The Pain Interference Score is the mean of these seven interference ratings, with a lower score being better.
Changes in health-related quality of life_ Eastern Cooperative Oncology Group score | approximately 36 weeks.
  To determine the impact of re-challenge 177Lu-PSMA-617 therapy on performance status using Eastern Cooperative Oncology Group score (ECOG) through re-challenge therapy completion. The ECOG Performance Status Scale is a widely used measurement in clinical oncology to assess a patient's level of functioning. It helps describe how a patient's disease impacts their daily living abilities. the ECOG scale ranges from 0 to 5. with a lower score indicating better daily living ability.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States